CLINICAL TRIAL: NCT04624997
Title: Evaluation de la COagulopathie et de la Dysfonction enDOthéliale Comme Facteur prédictif de la gravité de l'Infection Par SARS-CoV-2 / COVID-19
Brief Title: Coagulopathy and Vasculopathy Assessment as a Predictor of the Severity of SARS-CoV-2 / COVID-19 Infection
Acronym: SARCODO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: National Research Agency, France (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200521; 2020-A01048-31 (Other: Agence nationale de sécurité du médicament et des produits de santé (French Competent Authority))
Record Dates: First submitted 2020-06-17; First posted 2020-11-12 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: COVID-19; SARS-CoV-2 Infection
Keywords: COVID-19; SARS-CoV-2 infection; Hemostasis; Coagulopathy; Vasculopathy Assessment; Anticoagulant therapy
MeSH Terms: conditions — COVID-19; Hemostatic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, plasma, pellet
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient suspected COVID-19: Follow-up of patients as usual in care for infection. No specific puncture. Blood sample collect at admission and every 72h during hospitalisation for hemostasis evaluation, DNA extraction, Circulating endothelial cells measuring.
  Sampling can be delayed for 24h to match a planned blood collection for care or other research.
  Interventions: Other: biological sample

INTERVENTIONS:
Other: biological sample — biological sample

SUMMARY:
On 30 January 2020, WHO declared the SARS-CoV-2 outbreak as a public health emergency of international concern. Compared to SARS-CoV, which caused an outbreak of SARS in 2003, SARS-CoV-2 has a higher transmission capacity. Although the clinical manifestations of SARS-CoV-2 are dominated by respiratory symptoms, some patients have severe cardiovascular damage. In addition, patients with underlying cardiovascular disease may be at increased risk of death. Therefore, understanding the impairments caused by SARS-CoV-2 to the cardiovascular system and the underlying mechanisms is of the utmost importance.

Circulating endothelial cells (CECs) are generally considered markers of lesions and may be non-invasive markers of pulmonary vascular dysfunction during SARS-CoV-2 infection. Another marker of endothelial activation could be circulating extracellular vesicles. They could also be involved in the spread of the virus. Thus this project proposes to study different aspects of the diagnosis and pathophysiology of SARS-CoV-2. We propose to fully study activation state of coagulation and endothelium on a plasma and cellular side in patients diagnosed with SARS-CoV-2/COVID19. The different forms of the disease will be included: without lung disease, with a more or less severe lung disease, i.e. having evolved or not towards acute respiratory distress syndrome (ARDS). Extensive research of biomarkers will be compared to the detection of the virus in the respiratory tract as well as in the blood. This work will contribute to a better description of disease pathophysiology and should allow us to identify a patient profile in whom preventive or curative anticoagulant therapy could be considered.

DETAILED DESCRIPTION:
In December 2019, an outbreak of pneumonia caused by a new coronavirus occurred in Wuhan and spread rapidly throughout China, with the evolution towards a global pandemic. Originally called new coronavirus 2019 (2019-nCoV), the virus was later officially named Coronavirus 2 of Severe Acute Respiratory Syndrome (SARS-CoV-2) by WHO. On 30 January 2020, WHO declared the SARS-CoV-2 outbreak as a public health emergency of international concern. Compared to SARS-CoV, which caused an outbreak of SARS in 2003, SARS-CoV-2 has a higher transmission capacity. Although the clinical manifestations of SARS-CoV-2 are dominated by respiratory symptoms, some patients have severe cardiovascular damage. In addition, patients with underlying cardiovascular disease may be at increased risk of death. Therefore, understanding the impairments caused by SARS-CoV-2 to the cardiovascular system and the underlying mechanisms is of the utmost importance. During this Chinese epidemic, a coagulopathy was found in severe cases of SARS-CoV-2 infection, including significantly higher levels of D-dimers in severe forms, disturbed PT and aPTT ratio compared to survivors (P <0.05). 71.4% of non-survivors and 0.6% of survivors met the criteria for disseminated intravascular clotting during their hospital stay. This study was confirmed in a second Chinese population where DDimers are still correlated with mortality. The hypothesis of microthrombosis at the renal level was also associated with activation of coagulation since high levels of creatinine were associated with higher levels of DDimers, in favor of a thrombotic origin for kidney failure. Endothelial dysfunction may thus have a major role in the respiratory physiopathologic process as well as in the viral dissemination processes. Indeed, the SARS-CoV-2 receptor (ACE2) is strongly expressed in endothelial cells. Infection of endothelial cells could cause a lesion of the endothelium but also an activation that can trigger the activation of coagulation. Circulating endothelial cells (CECs) are generally considered markers of lesions and may be non-invasive markers of pulmonary vascular dysfunction during SARS-CoV-2 infection. Another marker of endothelial activation could be circulating extracellular vesicles. They could also be involved in the spread of the virus. Thus this project proposes to study different aspects of the diagnosis and pathophysiology of SARS-CoV-2. We propose to fully study activation state of coagulation and endothelium on a plasma and cellular side in patients diagnosed with SARS-CoV-2/COVID19. The different forms of the disease will be included: without lung disease, with a more or less severe lung disease, i.e. having evolved or not towards acute respiratory distress syndrome (ARDS). Extensive research of biomarkers will be compared to the detection of the virus in the respiratory tract as well as in the blood. This work will contribute to a better description of disease pathophysiology and should allow us to identify a patient profile in whom preventive or curative anticoagulant therapy could be considered.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years old
* Hospitalized for suspected COVID-19 in the medical wards or intensive care unit.
* Patients benefiting from a social security scheme
* Patient who has been informed of the study

Exclusion Criteria:

* Patients under guardianship / curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Public hospital patients
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-06-08 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Measure D-dimers (ng/ml) to study coagulopathy to characterize COVID-19 | 28 days
  Characterize COVID-19 and identify patient populations who will develop or aggravate a micro or macro thrombotic process
Measure fibrin monomers (µg/ml) to study coagulopathy to characterize COVID-19 | 28 days
  Characterize COVID-19 and identify patient populations who will develop or aggravate a micro or macro thrombotic process

SECONDARY OUTCOMES:
Study troponin (ng/ml) to characterize COVID-19 and identify patient populations who will develop or aggravate a micro or macro thrombotic process | 28 days
Study von Willebrand factor antigen (%) to characterize COVID-19 and identify patient populations who will develop or aggravate a micro or macro thrombotic process | 28 days
Study association of genetical and constitutive factors of thrombophilia :blood type ABO and COVID-19 severity according to OMS classification | 28 days
Study association of genetical and constitutive factors of thrombophilia: deficit in S protein and COVID-19 severity according to OMS classification | 28 days
Study association of genetical and constitutive factors of thrombophilia:deficit in C protein and COVID-19 severity according to OMS classification | 28 days
Study association of genetical and constitutive factors of thrombophilia: mutation in V factor of coagulation and COVID-19 severity according to OMS classification | 28 days
Study association of genetical and constitutive factors of thrombophilia:mutation in II factor of coagulation and COVID-19 severity according to OMS classification | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: David M Smadja, Principal Investigator — HEGP, AP-HP
Locations (2):
- France (2):
  - Hôpital Cochin, Paris
  - Hôpital Européen Georges Pompidou, Paris

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in publication could be shared. IPD detailed in the protocol of a planned metaanalysis could be shared.
Supporting Information: Study Protocol, ICF
Time Frame: One year after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on scientific project and scientific involvement of the PI team. The founder could be involved in the decision.
  Teams wishing obtain IPD must meet the sponsor and IP team to present scientifics (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractualization.